CLINICAL TRIAL: NCT06279286
Title: A Randomized, Double-blind, Placebo-controlled Phase Ⅰb/Ⅱ Study to Investigate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-10506 in Chinese Adult Participants With Insomnia Disorder
Brief Title: Phase Ⅰb/Ⅱ Study of HS-10506 in Chinese Participants With Insomnia Disorder
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10506-201
Record Dates: First submitted 2024-02-18; First posted 2024-02-28 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-02

CONDITIONS: Insomnia Disorder
Keywords: Clinical trial; insomnia disorder; phase Ⅰb/Ⅱ
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HS-10506, 10 milligram (mg) and placebo (Experimental): Phase Ib part: Participants will receive either 10mg of HS-10506 or matching placebo at night on Day 1 up to Day 5. Phase II part: Participants will receive either 10mg of HS-10506 or matching placebo at night on Day 1 up to Day 28.
  Interventions: Drug: HS-10506; Drug: Placebo
- HS-10506, 20 milligram (mg) and placebo (Experimental): Phase Ib part: Participants will receive either 20mg of HS-10506 or matching placebo at night on Day 1 up to Day 5. Phase II part: Participants will receive either 20mg of HS-10506 or matching placebo at night on Day 1 up to Day 28.
  Interventions: Drug: HS-10506; Drug: Placebo
- HS-10506, 40 milligram (mg) and placebo (Experimental): Phase Ib part: Participants will receive either 40mg of HS-10506 or matching placebo at night on Day 1 up to Day 5. Phase II part: Participants will receive either 40mg of HS-10506 or matching placebo at night on Day 1 up to Day 28.
  Interventions: Drug: HS-10506; Drug: Placebo
- HS-10506, 80 milligram (mg) and placebo (Experimental): Phase Ib part: Participants will receive either 80mg of HS-10506 or matching placebo at night on Day 1 up to Day 5. Phase II part: Participants will receive either 80mg of HS-10506 or matching placebo at night on Day 1 up to Day 28.
  Interventions: Drug: HS-10506; Drug: Placebo

INTERVENTIONS:
Drug: HS-10506 — HS-10506, tablets (10mg, 20mg, 40mg and 80mg) at night once daily from Day 1 to Day 5 in phase Ib study, and from Day 1 to Day 28 in phase II study.
Drug: Placebo — Placebo, placebo tablets matching the HS-10506 tablets

SUMMARY:
The primary purpose of this phase Ⅰb/Ⅱ study is to investigate the safety, tolerability, pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time) after multiple dose administration and the efficacy of HS-10506 (change versus placebo) on latency to persistent sleep (LPS) measured by polysomnography (PSG) in Chinese adult participants with insomnia disorder.

DETAILED DESCRIPTION:
This study consists of two stages: phase Ib and phase II. Primary objective of phase Ib Study is to assess the safety, tolerability of HS-10506 in subjects with insomnia disorder. .

Primary objective of phase II Study is to assess the efficacy of HS-10506 in subjects with insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 to 64 years of age, inclusive
2. Subjects are required to voluntarily sign the informed consent form;
3. Body mass index (BMI): for phase Ib, males must weigh at least 50 kilogram (kg), females at least 45 kg, and BMI (weight/height2 [kg/m2]) must be in the range of 18 to 30 kg/m2 (inclusive) for both gender; for phase II, BMI must be in the range of 18 to 35 kg/m2 (inclusive);
4. Participant must meet Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) criteria for insomnia disorder;
5. Participants must have Insomnia Severity Index (ISI) scores >=15 at screening and baseline;
6. Subjective sleep assessment: for phase Ib, subjects must have a self-reported sleep latency (sSOL) >= 30 minutes, a subjective sleep awakening time (sWASO) >= 30 minutes, and a subjective total sleep time (sTST) =< 6.5 hours using the sleep diary for at least three nights every week in the last 1 month prior to screening; For phase II, subjects must have an sSOL >= 30 minutes, sWASO >= 30 minutes, and sTST =< 6.5 hours for at least three nights every week within one month prior to screening; and sSOL >= 30 minutes, sWASO >= 30 minutes, and sTST =< 6.5 hours for at least 3 nights from sleep diary in the last 7 days;
7. PSG: for phase Ib, participants must demonstrate an LPS >= 20 minutes, TST < 420 minutes, and WASO >= 30 minutes at screening; for phase II, participants must demonstrate a 2-night mean LPS >= 30 minutes with neither night < 20 minutes, a 2-night mean TST =< 6.5 hours with neither night > 7 hours and a 2-night mean WASO >= 30 minutes with neither nigh < 20 minutes.

Exclusion Criteria:

1. Has history of or current sleep-wake disorders or sleep-related breathing disorders other than insomnia disorder, such as restless legs syndrome, periodic limb movement disorder, circadian rhythm disorder, narcolepsy, rapid eye movement sleep phase (REM) behavioral disorders, and obstructive sleep apnea;
2. Has a hypopnea index (AHI) >10 times/hour or periodic leg movement index (PLMI) >10 times/hour monitored by PSG at screening or run-in period;
3. Has history of or current neurodevelopmental retardation, cognitive impairment, epilepsy, schizophrenia, bipolar disorder, hyperthyroidism, cancer, severe cardio-cerebrovascular diseases or respiratory diseases; or clinically significant and/or unstable neurological, psychiatric, respiratory, cardiovascular, digestive, immunologic, urologic, endocrine diseases within the past 3 months prior to screening; or other systemic diseases that are inappropriate for the study;
4. (For phase II only) Has a Hamilton Anxiety Scale (HAMA) score >= 14 or Hamilton Depression Scale (HAMD-17) score >= 18;
5. Use of any medication that may affect the pharmacokinetics of HS-10506 within the past 2 weeks or 5 half-lives of the medication;
6. Use of any medication that may affect sleep-wake function, or any other prohibited central nervous system active medications within 1 week or 5 half-lives of the medication;
7. Has received systemic hypnotherapy, cognitive behavioral therapy (CBT), or other non-pharmacological treatments for insomnia in last 4 weeks or have plans during the study;
8. Working across 3 or more time zones or shift work within 2 weeks prior to screening;
9. Regularly naps more than 3 naps per week for > 1 hour each time within the past 2 weeks prior to screening;
10. Has a risk of suicide according to the Columbia Suicide Severity Rating Scale (C-SSRS), or has a high risk of suicide at the discretion of the investigator;
11. Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 312 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE) | Baseline up to the end of the study (3 days after the last dose) or early withdrawal
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Incidence and severity of serious adverse events (SAE) | Baseline up to the end of the study (3 days after the last dose) or early withdrawal
  An SAE is any adverse event (AE) that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Changes in laboratory test before and after drug administration | Baseline up to the end of the study (3 days after last dose) or early withdrawal
  Number of participants with clinically significant laboratory abnormalities, including complete blood cell count, urinalysis, serum chemistry, coagulation function were reported.
Changes in ECG before and after drug administration | Baseline up to the end of the study (3 days after last dose) or early withdrawal
  Number of participants with clinically significant ECG abnormalities were reported.
Changes in Karolinska Sleepiness Scale (KSS) scores before and after drug administration | From start of the drug administration to the next day of the last dose or early withdrawal
  The KSS is a patient-reported assessment of drowsiness level at the time of scale administration.
Change from baseline in the mean LPS measured by PSG on Night 13 and Night 14 | Baseline, Night 13& Night 14
  LPS is the time in minutes from 'lights out' that marks the starting of total recording time to the first epoch recorded as sleep.

SECONDARY OUTCOMES:
The maximum plasma concentration (C[max]) | Baseline up to 48 hours after the last dose or early withdrawal
  The C[max] is the maximum observed plasma concentration and will be determined for HS-10506.
Time to reach the maximum plasma concentration (T[max]) | Baseline up to 48 hours after the last dose or early withdrawal
  Time to reach maximum observed plasma concentration (T[max]) of HS-10506.
Area under the plasma concentration-time curve from time zero to last time of quantifiable concentration (AUC[0-t]) | Baseline up to 48 hours after the last dose or early withdrawal
  Area under the concentration-time curve from time zero to last time of quantifiable concentration of HS-10506.
Terminal elimination half-life (t1/2) | Baseline up to 48 hours after the last dose or early withdrawal
  Apparent terminal elimination half-life of HS-10506.
Change in latency to persistent sleep (LPS) relative to baseline on night 5 of PSG monitoring | Baseline and Night 5
  Latency to persistent sleep (LPS) is the time in minutes from 'lights out' that marks the starting of total recording time to the first epoch recorded as sleep over PSG assessment.
Change in Wake After Sleep Onset (WASO) relative to baseline on night 5 of PSG monitoring | Baseline and Night 5
  Wake After Sleep Onset (WASO) is defined as the duration of wakefulness from the onset of persistent sleep over the PSG assessment.
Change from baseline in mean LPS measured by PSG | Baseline up to 28 days.
  Latency to Persistent Sleep (LPS) is the time in minutes from 'lights out' that marks the starting of total recording time to the first epoch recorded as sleep over PSG assessment.
Change from baseline in mean TST measured by PSG | Baseline up to 28 days.
  Total sleep time (TST) is the total amount of sleep time scored during the total recording time over PSG assessment.
Change from baseline in mean WASO measured by PSG | Baseline up to 28 days.
  Wake after initial sleep onset (WASO) is defined as the duration of wakefulness from the onset of persistent sleep over PSG assessment.
Change from baseline in the mean values of self-reported sleep-onset latency (sSOL) recorded in the sleep diary | Baseline up to 28 days.
  Change from baseline in the mean values of self-reported sleep-onset latency (sSOL) measured by sleep diary.
Change from baseline in the mean values of self-reported total sleep time (sTST) recorded in the sleep diary | Baseline up to 28 days.
  Change from baseline in mean self-reported total sleep time measured by sleep diary.
Incidence and severity of adverse events (AE) | Baseline up to 28 days.
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Incidence and severity of serious adverse events (SAE) | Baseline up to 28 days.
  An SAE is any adverse event (AE) that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China